CLINICAL TRIAL: NCT03767686
Title: Covered Endovascular Reconstruction of Aortic Bifurcation (CERAB) for Extensive Aortoiliac Occlusive Disease A Multicenter, Prospective Investigator Initiated Trial
Brief Title: Covered Endovascular Reconstruction of Aortic Bifurcation (CERAB) for Extensive Aortoiliac Occlusive Disease
Status: Terminated | Type: Observational
Why Stopped: Finance stop
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, Principal Investigator, Rijnstate Hospital
Other Study IDs: CERAB trial
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Aorto-Iliac Atherosclerosis; Aortoiliac Obstruction
MeSH Terms: conditions — Leriche Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endovascular treatment is rapidly taking over surgery for aorto-iliac occlusive disease (AOID), also in extensive pathology. This is related to its minimally invasiveness, decreasing the procedural morbidity rate. When the aortic bifurcation was involved in the lesion, the patency rates of kissing stents configurations were often inferior to open repair. In 2013 the Covered Endovascular Reconstruction of the Aortic Bifurcation (CERAB) technique was introduced in an attempt to improve endovascular treatment results by a more anatomical and physiological reconstruction, with a subsequent improved clinical outcome.

This investigator-initiated multicenter trial will prospectively record all data on performed CERAB procedures using the Bentley balloon expandable covered stents (BeGraft Aortic and BeGraft Peripheral) in multiple International sites, in order to gain more robust real-world data on the efficacy of these stent grafts for this indication.

Consecutive patients in whom a CERAB will be performed with these particular covered stents in the participating centers.

Main study parameters/endpoints: The primary end-point of this study is technical success. Patency rates, peri-procedural morbidity, clinical improvement, quality of life, clinically-driven target vessel revascularization and reintervention-rate will be secondary outcome measures. Overall, patients will be followed for 5 years

DETAILED DESCRIPTION:
Endovascular treatment is rapidly taking over surgery for aorto-iliac occlusive disease (AOID) also for complex lesions. This is related to the minimally invasiveness of the procedure decreasing the morbidity rate. Patency results of endovascular treatment were often inferior compared to open repair when the aortic bifurcation was involved in the lesion. In 2013 Covered Endovascular Reconstruction of the Aortic Bifurcation (CERAB) technique was introduced in an attempt to improve endovascular treatment results by a more anatomical and physiological reconstruction, with a subsequent better clinical outcome. The early results of the CERAB configuration are promising with primary, primary-assisted and secondary patency of, respectively 86.2%/91.1%/97.0% at 1-year, 83.9%/88.7%/97.0% at 2-year and 82.1%/86.8%/97.0% at 3-year FU in a group of 130 patients, including the first in man results. The vast majority (89.2%) were TASC-II D lesions and the 30-day major complication rate was 7.7%.

This trial is designed to prospectively collect all data on implanted CERAB configurations, using the balloon expandable stents from Bentley InnoMed, in a defined group of aorto-iliac pathology in multiple international sites in order to gain more insight in the outcome of the technique. Technical success will be the primary endpoint. Other evaluations will include patency rates, quality of life, the reintervention-rate, 30-day morbidity and target vessel revascularization up to 5 years after treatment.

A total of 145 patients will be included and followed until 5 years of follow-up. A core lab will independently analyze the images (CT scan or duplex) which will be made at the following time points: pre-op, 1 month, 6 months, 1 year and yearly up to 5 years of follow-up.

Additionally, at these time points three questionnaires will be completed by the patients. These questionnaires are about walking ability (WIQ), and quality of life (EQ-5D and WHOQoL-BREF).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Provided written informed consent
* Clinical necessity for treatment
* Eligible anatomy for CERAB without the need for chimney's
* TASC-2 classification as assigned in the study protocol (specified type B, C and D lesions)

Exclusion Criteria:

* Patient is participating in another conflicting clinical study
* Patient's life expectancy <2 years as judged by the investigator
* Patient has a psychiatric or other condition that may interfere with the study
* Patient has a known allergy to any device component
* Patients with a systemic infection who may be at increased risk of endovascular graft infection.
* Patient has a coagulopathy or uncontrolled bleeding disorder
* Patient had a CVA or an MI within the prior three months
* Patient is pregnant (Female patients of childbearing potential only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 145 patients in whom a CERAB will be performed.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Technical success | Up to 30 days
  Technical success is defined as successful implantation of the CERAB device without occlusion during the first 30-days after implantation
Primary patency | Up to 12 months
  Primary patency at 12 months measured by duplex ultrasound
Technical success | Up to 30 days
  Technical success is defined as successful implantation of the CERAB device without conversion to open repair

SECONDARY OUTCOMES:
Technical success | Up to 5 years of follow-up
  Patency rates measured by duplex ultrasound
Technical success | Up to 5 years of follow-up
  Target vessel revascularization measured by duplex ultrasound
Technical success | Up to 5 years of follow-up
  Conversion to open surgery judged at every clinic visit by the investigator
Clinical success | Up to 5 years of follow-up
  Freedom from reinterventions judged at every clinic visit by the investigator
Clinical success | Up to 30 days of follow-up
  30 days morbidity judged at every clinic visit by the investigator
Clinical success | Up to 3 months of follow-up
  Incidence serious adverse events device related judged at every clinic visit and in between visits if the investigator notes that an AE appeared, done by the investigator
Clinical success | Up to 6 months of follow-up
  Incidence serious adverse events device related judged at every clinic visit and in between visits if the investigator notes that an AE appeared, done by the investigator
Clinical success | Up to 12 months of follow-up
  Incidence serious adverse events device related judged at every clinic visit and in between visits if the investigator notes that an AE appeared, done by the investigator
Clinical success | Up to 3 months of follow-up
  Incidence of serious adverse events procedure related judged at every clinic visit and in between visits if the investigator notes that an AE appeared, done by the investigator
Clinical success | Up to 6 months of follow-up
  Incidence of serious adverse events procedure related judged at every clinic visit and in between visits if the investigator notes that an AE appeared, done by the investigator
Clinical success | Up to 12 months of follow-up
  Incidence of serious adverse events procedure related judged at every clinic visit and in between visits if the investigator notes that an AE appeared, done by the investigator
Clinical success | Up to 5 years of follow-up
  Overall survival investigated with every clinic visit, done by the investigator
Clinical success | Up to 5 years of follow-up
  Reintervention-free survival investigated with every clinic visit, done by the investigator
Clinical success | Up to 5 years of follow-up
  Clinical improvement as measured by the Rutherford category of which 1 is better dan 6
Clinical success | Up to 5 years of follow-up
  Patient reported outcomes measured by the EQ-5D questionnaire
Clinical success | Up to 5 years of follow-up
  Patient reported outcomes measured by the Walking Impairment Questionnaire
Clinical success | Up to 5 years of follow-up
  Patient reported outcomes measured by the WHOQoL Bref

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, PhD, Principal Investigator — Principal Investigator
Locations (8):
- Dandenong Hospital, Victoria Point, Australia
- A.O.U. Città della Salute e della Scienza di Torino, Torino, Italy
- Spanish Hospital, Mexico City, Mexico
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Dijklander Ziekenhuis, Hoorn
  - Medical University Center Maastricht, Maastricht
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton